CLINICAL TRIAL: NCT01497964
Title: A Phase 2, Multicenter Study of Cabazitaxel Single Agent Administered as a 1-Hour Intravenous Infusion Every 3 Weeks to Evaluate the Safety, Tolerability and Anti-tumor Activity of Cabazitaxel in Patients With Advanced Gastric Adenocarcinoma Who Have Failed Prior Chemotherapy Regimens
Brief Title: Cabazitaxel in Asian Patients With Advanced Gastric Cancer Who Failed Prior Chemotherapy
Acronym: GASTANA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD12417; U1111-1121-6247 (Other: UTN)
Record Dates: First submitted 2011-12-06; First posted 2011-12-23 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel, several dosages
  Interventions: Drug: cabazitaxel XRP6258

INTERVENTIONS:
Drug: cabazitaxel XRP6258 — Pharmaceutical form: solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

- To evaluate the anti-tumor activity of cabazitaxel by assessing objective tumor response rate (ORR) at the recommended dose (RD) when administered as a single agent every 3 weeks in patients with advanced gastric adenocarcinoma who have failed prior chemotherapy regimens

Secondary Objectives:

* To determine the RD of cabazitaxel when administered as a single agent every 3 weeks
* To evaluate safety of cabazitaxel when administered as a single agent every 3 weeks
* To estimate the overall survival (OS) and progression free survival (PFS)
* To assess the pharmacokinetics (PK) profile of cabazitaxel in part 1

DETAILED DESCRIPTION:
Patients will be treated until disease progression, unacceptable toxicity, or patient's refusal of further study treatment. All patients will be followed during and after the study treatment until death or the end of study, whichever comes first.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed unresectable or metastatic gastric adenocarcinoma including adenocarcinoma of gastroesophageal junction, which have failed 2 prior chemotherapy regimens. (For countries where a standard of care has not been established for the 2nd line treatment for advanced gastric cancer, those who failed 1 or 2 prior chemotherapy regimens can be included)
* Signed informed consent

Exclusion criteria:

* Patients who have received >2 prior systemic chemotherapy regimens for advanced gastric cancer.
* For patients entering part 2, those without at least one measurable lesion at baseline according to Response Evaluation Criteria in Solid Tumors 1.1 criteria
* Eastern Cooperative Oncology Group performance status >1
* Age <18 years
* Inadequate organ and bone marrow function
* Prior surgery, chemotherapy, targeted agents, investigational agents, or other anti-cancer therapy within 4 weeks prior to enrollment in the study
* Prior radiation therapy within 6 weeks prior to enrollment (except palliative radiation for a local pain control)
* Previous treatment with cabazitaxel
* Known brain or leptomeningeal involvement of cancer
* Patients with known acquired immunodeficiency syndrome (AIDS) related illness or known HIV infection requiring antiretroviral treatment.
* Patients with active varicella zoster infection, or known hepatitis B or C infection.
* History of severe hypersensitivity reaction ≥ grade 3 to drugs formulated with polysorbate 80 such as docetaxel

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to a maximum of 2 years
Progression free survival (PFS) | Up to a maximum of 2 years
Number of patients with adverse events | Up to a maximum of 2 years
Pharmacokinetic parameter: Cmax | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion..
Pharmacokinetic parameter tmax | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion..
Pharmacokinetic parameter t1/2z | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion..
Pharmacokinetic parameter AUC | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion
Pharmacokinetic parameter AUClast | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion
Pharmacokinetic parameter CL | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion
Pharmacokinetic parameter Vss | pre-infusion, end of infusion, 5, 15, 30 min, 1, 3, 5, 8 hours after end of infusion, 24, 48, 72, 120, 168, 216 hours after start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 410001, Seoul, South Korea